CLINICAL TRIAL: NCT05493488
Title: An Observer-Blinded, Randomized, Aqueous Gel Controlled Trial of the Safety and Efficacy of DBI-001 Gel, DBI-002 Gel, and Aqueous Gel in Subjects With Interdigital Tinea Pedis
Brief Title: A Trial to Evaluate the Safety and Efficacy of DBI-001 Gel, DBI-002 Gel, and Aqueous Gel in Subjects With Tinea Pedis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-210
Record Dates: First submitted 2022-07-26; First posted 2022-08-09 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-09

CONDITIONS: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — BANG polymer gel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DBI-001 Gel (Active Comparator): Topical application of DBI-001 Gel on foot/feet affected with tinea pedis
  Interventions: Biological: DBI-001 Gel
- DBI-002 Gel (Active Comparator): Topical application of DBI-002 Gel on foot/feet affected with tinea pedis
  Interventions: Biological: DBI-002 Gel
- Aqueous Gel (Placebo Comparator): Topical application of Aqueous Gel on foot/feet affected with tinea pedis
  Interventions: Biological: Aqueous Gel

INTERVENTIONS:
Biological: DBI-001 Gel — Topical application of DBI-001 gel on foot/feet affected with tinea pedis
  Arms: DBI-001 Gel
Biological: DBI-002 Gel — Topical application of DBI-002 gel on foot/feet affected with tinea pedis
  Arms: DBI-002 Gel
Biological: Aqueous Gel — Topical application of Aqueous gel on foot/feet affected with tinea pedis
  Arms: Aqueous Gel

SUMMARY:
This is a randomized, observer blinded, Aqueous Gel-controlled trial examining the effect of daily application for approximately 6-8 days of DBI-001 Gel, DBI-002 Gel, and Aqueous Gel on the subjects with interdigital tinea pedis based on Whole Genome Sequencing (WGS) and Quantitative Polymerase Chain Reaction (qPCR), and comparison between Quantitative Polymerase Chain Reaction (qPCR) and Potassium Hydroxide (KOH) for the presence of Trichophyton rubrum (T.rubrum) as well as signs and symptoms and local tolerability and toxicity on treated sites in subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand, agree to, and sign the study Informed Consent
2. A signed Health Information Portability and Accountability Act (HIPAA) authorization form which permits the use and disclosure of the subject's individually identifiable health information.
3. Male or Female Subjects of any race 18-65 years of age.
4. Subjects with a clinical diagnosis of interdigital T. pedis.
5. Investigator confirmed diagnosis by a positive T. rubrum potassium hydroxide (KOH) wet mount at Screening at the investigative site.
6. A quantifiable level of T. rubrum based on Sponsor laboratory qPCR from the sample obtained at the Screening visit.
7. The sum of the clinical signs and symptoms scores of at least one web space (Target web space) is at least 4 using the Grading of Signs and Symptoms of T. pedis including a minimum score of 2 for erythema AND a minimum score of 2 for either scaling/fissures or pruritus/burning (on a scale of 0-3, where 2 indicates moderate severity).
8. Target web space(s) should have an adequate amount of leading-edge scale to provide enough scale sampling for KOH.

Exclusion Criteria:

1. Women who are pregnant, planning a pregnancy, breastfeeding or have a positive pregnancy test at screening.
2. Any dermatological conditions that could interfere with clinical evaluations
3. The clinical diagnosis of moccasin T. pedis.
4. Subjects with gram negative interdigital tinea pedis based on a clinical diagnosis: Gram-negative athlete's foot - the interspace is foul smelling, whitish, painful, strongly macerated, and hyperkeratotic with erosions, exudation, and intense inflammation and often disabling.
5. Any underlying disease(s) or other dermatological condition that requires the use of interfering topical or systemic therapy.
6. Subjects with concurrent use of any of the following topical preparations who have not completed the specified washout period(s) for the following topical medications applied to the foot at the time of the Screening visit:

   1. Washout of 1 week prior to the screening visit for topical astringents and abrasives (e.g., Burrow's solution), Vicks VapoRub, tea tree oil)
   2. Washout of 2 weeks prior to the screening visit for topical antibiotics and antifungal on the feet (e.g., Neomycin, Miconazole, Clotrimazole, Terbinafine)
   3. Washout of 4 weeks prior to the screening visit for the topical Anti-inflammatories, corticosteroids, topical immunomodulators on the feet (e.g., Pimecrolimus, Tacrolimus)
7. Subjects with concurrent use of any of the following systemic medications who have not completed the specified washout period(s) for the following systemic medications at the time of the Screening visit:

   1. Washout of 4 weeks prior to the screening visit for the systemic corticosteroids (including intramuscular injections) (e.g., Triamcinolone acetonide)
   2. Washout of 4 weeks prior to the screening visit for the systemic antibiotics (e.g., Tetracycline, Cephalosporins, etc.) and/or Antifungal agents (e.g., Fluconazole, Itraconazole, Terbinafine, etc.)
   3. Washout of 4 weeks prior to the screening visit for the systemic immunomodulators (e.g., Cyclophosphamide, Azathioprine, Biologicals-Monoclonal Antibodies)
8. Treatment of any type of cancer within the last 6 months except for superficial skin cancers such as basal cell carcinoma and squamous cell carcinoma.
9. History of any significant internal disease which contraindicates use of a live microbiome (e.g., leukemia, liver failure, cardiovascular disease).
10. Subjects who are known to be allergic to any of the Test article(s) or any components in the test article(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
11. AIDS or AIDS related complex by medical history.
12. History of current street drug or alcohol abuse, or street drug or alcohol abuse within the past year.
13. Known or suspected immune suppressive medications or diseases.
14. Subjects with poorly controlled diabetes mellitus Type I or II requiring medical intervention/treatment.
15. Peripheral vascular disease based on medical history.
16. Any subject not able to meet the study attendance requirements.
17. Subjects who have participated in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.
18. Use of any orthopedic appliance (e.g., cast, soft cast, splint) on either foot or ankle, or surgery of either foot or ankle within 90 days of the Screening visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in abundance of T. rubrum based on Quantitative Polymerase Chain Reaction (qPCR) | 14 days of participation
  Change in abundance of T. rubrum at baseline, day 7 and day 14

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | 14 days of participation
  Safety
Changes in signs and symptoms of T. Pedis | 14 days of participation
  Change from baseline in individual signs and symptoms of Tinea Pedis at days 7 and 14 of sites treated with DBI-001 Gel, DBI-002 Gel, or Aqueous Gel. The minimum value is 0 and the maximum value is 3 the subject's self reported observation on local tolerability.
Changes in the signs and symptoms and Investigators Static Global Assessment (ISGA) of Tinea Pedis | 14 days of participation
  Changes from Baseline in signs and symptoms and ISGA at Days 7 and 14
Change in abundance of T. rubrum based on qPCR and WGS | 14 days of participation
  Antimicrobial efficacy
Molecular diagnostic qPCR and WGS comparison of DBI-001 Gel, DBI-002 Gel and Aqueous Gel | 14 days of participation
  Antimicrobial efficacy and microbiome community analysis
Bacterial culture comparison of DBI-001 Gel, DBI-002 Gel and Aqueous Gel | 14 days of participation
  Antimicrobial efficacy and microbiome community analysis
Increase or decrease of colony forming units after DBI-001 Gel, DBI-002 Gel application | 14 days of participation
  Antimicrobial efficacy
Correlation between levels of DBI-001 Gel, DBI-002 Gel and abundance of T. rubrum based on qPCR | 14 days of participation
  Antimicrobial efficacy
Correlation between qPCR quantification and KOH for presence of T. rubrum at screening | 28 days from screening
  Compare sensitivity and specificity of qPCR analysis and KOH for presence of T. rubrum at Screening

CONTACTS AND LOCATIONS:
Overall Officials: Emma Taylor, Ph.D, Study Director — DermBiont, Inc.
Locations (2):
- United States (2):
  - Oregon Dermatology and Research, Portland, Oregon
  - Premier Clinical Research, Spokane, Washington